CLINICAL TRIAL: NCT05387122
Title: The Effect of Mandibular Advancement Devices on Markers of Cardiovascular Health in Mild to Moderate Obstructive Sleep Apnea Patients Who Are Non-Compliant With Continuous Positive Airway Pressure Therapy
Brief Title: The Effect of Mandibular Advancement Devices on Markers of Cardiovascular Health in Obstructive Sleep Apnea Patients
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108618
Record Dates: First submitted 2022-03-29; First posted 2022-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mandibular advancement device (MAD) — mandibular advancement device (MAD) is a removable oral appliance. It is an alternative therapy for patients of Obstructive Sleep Apnea who are non compliant to Continuous positive airway pressure(CPAP) which is the most accepted therapy for Obstructive Sleep Apnea.

SUMMARY:
Obstructive sleep apnea (OSA) is a type of disordered breathing defined by the repetitive obstruction of airflow during sleep due to upper airway collapse. Each obstructive event contributes to decreased blood oxygen, or hypoxia. OSA has been associated with various cardiovascular diseases, including hypertension, stroke, heart failure, and coronary artery disease. A factor in this association may be the decrease in blood vessel health and the marked over activation of the sympathetic nervous system that is observed in OSA due to nighttime hypoxia. The sympathetic nervous system is responsible for maintaining heart and blood vessel (cardiovascular) balance. Elevated sympathetic nervous activity (SNA) is a likely cause of hypertension and subsequent cardiovascular disease.

Continuous positive airway pressure (CPAP) therapy is the most accepted treatment for OSA and has been shown to improve high blood pressure and SNA in patients. An alternative therapy for OSA is a type of removable oral appliance known as a mandibular advancement device (MAD). Currently, there is no research directly measuring SNA in OSA patients using MADs. In addition to other cardiovascular markers, the investigators would like to directly assess SNA during a MAD intervention using the gold standard technique of microneurography. The investigators believe this will provide important information for the management of OSA, as levels of SNA are known to respond to both acute and chronic levels of hypoxia. Improved heart and blood vessel markers could further support MAD use, providing an important alternative therapy for those that can not tolerate CPAP.

DETAILED DESCRIPTION:
In OSA the obstruction of breathing can be either partial (hypopnea) or complete (apnea), and each obstructive event contributes to decreased blood oxygen, or hypoxia. Sleep disordered breathing and nighttime hypoxia have both been identified as independent risk factors of death. Specifically, OSA is estimated to affect 34% of men and 17% of women and when inadequately treated patients present with daytime sleepiness, depression, workplace accidents and cardiovascular disease.

The severity of OSA is determined by the apnea-hypopnea index (AHI) which is the average number of airway obstructions experienced per hour of sleep. CPAP therapy has been shown to improve high blood pressure, AHI and SNA in patients. However, benefits of CPAP therapy are dose-dependent and are largely affected by patient compliance. Unfortunately, due to various discomforts associated with the use of CPAP therapy, less than fifty percent of patients adhere to long-term therapy.

MADs have increased compliance in comparison to CPAP, and improve some patient's symptoms of sleepiness. Yet, MAD interventions have shown smaller improvements in AHI values when compared to CPAP. However, AHI has been criticized for being an overly simplistic measurement of nocturnal hypoxia. In contrast, SNA is known to respond both acutely and chronically to varying levels of blood oxygen. Therefore, MAD interventions may not produce changes in AHI equal to that of a CPAP intervention; however, they may change levels of SNA and other specific CV markers of blood vessel health. This would further support the use of MADs and provide additional insight into the underlying cardiovascular mechanisms involved in OSA therapy. Understanding and validating additional therapies for OSA is of great importance, due to the significant health consequences of the disease.

Objectives

The proposed investigation aims to determine the following in mild to moderate OSA patients who fail to comply with CPAP therapy:

Does MAD therapy improve AHI in mild to moderate severity OSA?

Does MAD therapy lower basal SNA in mild to moderate severity OSA?

Does MAD therapy improve vascular function, blood pressure, heart rate variability and blood markers of elevated SNA in mild to moderate severity OSA?

Research Method/ Procedures

Methodology

To address this hypothesis, the investigators propose a prospective case series examining subjects at baseline, at 3 months and again at 6 months after a MAD intervention. A 2020 study by Ruzicka et al. found no changes in SNA after a CPAP intervention of 6 weeks. Another study by Henderson et al, 2016, found a significant reduction in SNA during a CPAP intervention of 6 months and 12 months. In 2009, Kuramoto et al measured changes in SNA indirectly during a 3 month CPAP intervention and did not see significant results. Our methodology involves direct measurement of SNA during MAD therapy, therefore, testing intervals at baseline, 3 months and 6 months of MAD therapy have been selected.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-70
* Diagnosed with Obstructive Sleep Apnea and prescribed with Mandibular Advancement Device
* No medical history of cardiovascular, pulmonary, renal diseases

Exclusion Criteria:

* Any known cardiovascular, respiratory or pulmonary disease
* Have a history of smoking regularly in past 6 months
* Pre-existing symptomatic non-respiratory sleep disorder (restless leg syndrome, chronic insomnia)
* if more than 50% of their observed apneas are due to sleep apnea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers with mild to moderate OSA will be recruited with the assistance of referring dentists who are certified to provide MADs under the Alberta Dental Association & College guidelines. Participants will be included if they are between the ages of 18-70 years, initiating adjustable MAD therapy with their provider and no medical history of heart failure, cardiopulmonary and renal disease
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Difference in Sympathetic Nerve Activity | 3 months
  Muscle sympathetic nerve activity. Direct multi-unit postganglionic muscle sympathetic nerve activity (MSNA) will be obtained via microneurography. A sterile Tungsten recording microelectrode (35 mm long, 200 μm in diameter, tapered to a 1- to 5-μm uninsulated tip) will be inserted into a muscle nerve fascicle of a sympathetic nerve bundle, of the peroneal nerve. A reference electrode will also be inserted subcutaneously 1-3 cm from the recording electrode. MSNA will be obtained by manually manipulating the microelectrode until a characteristic bursting pattern is observed A trained researcher will record and analyze to quantify sympathetic activity as: burst frequency (bursts/min), burst incidence (bursts/ 100 heart beats), burst amplitude (normalized to largest resting amplitude), and total activity (burst frequency multiplied by mean normalized burst amplitude)
Difference in Cardiovascular markers - Heart Rate | 3 months
  All cardiovascular parameters will be acquired using an analog-to-digital converter (Powerlab/16SP ML 880; ADInstruments, Colorado Springs, CO, USA) interfaced with a personal computer. Commercially available software will be used to analyze ventilatory and cardiovascular variables (LabChart V7.1, ADinstruments, Colorado Springs, CO, USA). Throughout all procedures, heart rate will be determined from a standard lead III electrocardiogram (ML 132, ADInstruments, Colorado Springs, CO, USA). Heart Rate will be recorded in beats/ minute
Difference in Cardiovascular markers- Blood Pressure | 3 months
  All cardiovascular parameters will be acquired using an analog-to-digital converter (Powerlab/16SP ML 880; ADInstruments, Colorado Springs, CO, USA) interfaced with a personal computer. Commercially available software will be used to analyze ventilatory and cardiovascular variables (LabChart V7.1, ADinstruments, Colorado Springs, CO, USA). Throughout all procedures, Blood pressure will be recorded beat-by-beat by finger pulse photoplethysmograph; mmHg.
Fasted blood sample- Neurotransmitters | 3 months
  Fasted blood samples (~30ml) will be analyzed for sympathetic nervous system neurotransmitters (Norepinephrine, Epinephrine,)
Fasted blood sample- Sex Hormones | 3 months
  Fasted blood samples (~30ml) will be analyzed for sex hormones (estrogen, progesterone, testosterone)
Endothelial function- time to peak dilation | 3 months
  Flow Mediated Dilation: This will be assessed in the brachial artery, using an ultrasound system. A sphygmomanometer cuff will be placed and inflated around the forearm to a supra-systolic pressure (250 mmHg) to occlude forearm blood flow for 5 min. After this time period, the cuff will be rapidly deflated (~1 s). Baseline brachial artery blood flow velocity and diameter will be recorded for 1 minute before cuff inflation, and for 3.5 min beginning 30 s prior to cuff release. (FMD, time to maximal dilation; s)
Endothelial function- Flow mediated dilation | 3 months
  Flow Mediated Dilation: This will be assessed in the brachial artery, using an ultrasound system. A sphygmomanometer cuff will be placed and inflated around the forearm to a supra-systolic pressure (250 mmHg) to occlude forearm blood flow for 5 min. After this time period, the cuff will be rapidly deflated (~1 s). Baseline brachial artery blood flow velocity and diameter will be recorded for 1 minute before cuff inflation, and for 3.5 min beginning 30 s prior to cuff release. Percent change in artery diameter will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F Mir, DSc, Principal Investigator — University of Alberta; Craig Steinback, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. J Clin Invest. 1995 Oct;96(4):1897-904. doi: 10.1172/JCI118235. PMID 7560081
- [Background] Henderson LA, Fatouleh RH, Lundblad LC, McKenzie DK, Macefield VG. Effects of 12 Months Continuous Positive Airway Pressure on Sympathetic Activity Related Brainstem Function and Structure in Obstructive Sleep Apnea. Front Neurosci. 2016 Mar 10;10:90. doi: 10.3389/fnins.2016.00090. eCollection 2016. PMID 27013952
- [Result] de Vries GE, Wijkstra PJ, Houwerzijl EJ, Kerstjens HAM, Hoekema A. Cardiovascular effects of oral appliance therapy in obstructive sleep apnea: A systematic review and meta-analysis. Sleep Med Rev. 2018 Aug;40:55-68. doi: 10.1016/j.smrv.2017.10.004. Epub 2017 Oct 26. PMID 29195726
- [Result] Ferguson KA, Cartwright R, Rogers R, Schmidt-Nowara W. Oral appliances for snoring and obstructive sleep apnea: a review. Sleep. 2006 Feb;29(2):244-62. doi: 10.1093/sleep/29.2.244. PMID 16494093
- [Result] Imes CC, Baniak LM, Choi J, Luyster FS, Morris JL, Ren D, Chasens ER. Correlates of Endothelial Function in Older Adults With Untreated Obstructive Sleep Apnea and Cardiovascular Disease. J Cardiovasc Nurs. 2019 Jan/Feb;34(1):E1-E7. doi: 10.1097/JCN.0000000000000536. PMID 30303893
- [Result] Lopez-Jimenez F, Sert Kuniyoshi FH, Gami A, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. Chest. 2008 Mar;133(3):793-804. doi: 10.1378/chest.07-0800. No abstract available. PMID 18321908
- [Result] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Result] Meah VL, Busch SA, Jones KE, Davenport MH, Steinback CD. A review of acute responses, after-effects and chronic complications related to microneurography. Clin Neurophysiol. 2019 Oct;130(10):1781-1788. doi: 10.1016/j.clinph.2019.06.228. Epub 2019 Jul 15. PMID 31401486
- [Result] Ning Y, Zhang TS, Wen WW, Li K, Yang YX, Qin YW, Zhang HN, Du YH, Li LY, Yang S, Yang YY, Zhu MM, Jiao XL, Zhang Y, Zhang M, Wei YX. Effects of continuous positive airway pressure on cardiovascular biomarkers in patients with obstructive sleep apnea: a meta-analysis of randomized controlled trials. Sleep Breath. 2019 Mar;23(1):77-86. doi: 10.1007/s11325-018-1662-2. Epub 2018 Apr 22. PMID 29682699
- [Result] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Result] Phillips CL, Grunstein RR, Darendeliler MA, Mihailidou AS, Srinivasan VK, Yee BJ, Marks GB, Cistulli PA. Health outcomes of continuous positive airway pressure versus oral appliance treatment for obstructive sleep apnea: a randomized controlled trial. Am J Respir Crit Care Med. 2013 Apr 15;187(8):879-87. doi: 10.1164/rccm.201212-2223OC. PMID 23413266
- [Result] Punjabi NM, Caffo BS, Goodwin JL, Gottlieb DJ, Newman AB, O'Connor GT, Rapoport DM, Redline S, Resnick HE, Robbins JA, Shahar E, Unruh ML, Samet JM. Sleep-disordered breathing and mortality: a prospective cohort study. PLoS Med. 2009 Aug;6(8):e1000132. doi: 10.1371/journal.pmed.1000132. Epub 2009 Aug 18. PMID 19688045
- [Result] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Result] Zinchuk A, Yaggi HK. Phenotypic Subtypes of OSA: A Challenge and Opportunity for Precision Medicine. Chest. 2020 Feb;157(2):403-420. doi: 10.1016/j.chest.2019.09.002. Epub 2019 Sep 17. PMID 31539538
- [Result] Yamamoto U, Nishizaka M, Tsuda H, Tsutsui H, Ando SI. Crossover comparison between CPAP and mandibular advancement device with adherence monitor about the effects on endothelial function, blood pressure and symptoms in patients with obstructive sleep apnea. Heart Vessels. 2019 Oct;34(10):1692-1702. doi: 10.1007/s00380-019-01392-3. Epub 2019 Mar 29. PMID 30927057